CLINICAL TRIAL: NCT06609434
Title: The Role and Safety of Radiofrequency Ablation in the Multidisciplinary Treatment of Intrahepatic Recurrence After Colorectal Cancer Liver Metastasis Surgery
Brief Title: The Role and Safety of Radiofrequency Ablation in Recurrent Liver Metastasis of Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2-2157
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Colo-rectal Cancer; Liver Metastasis
Keywords: Colo-rectal cancer; Liver Metastasis; radiofrequency ablation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: The study was divided into two groups, the interventional group was: systemic therapy combined with radiofrequency therapy, the control group was: systemic therapy alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic therapy (No Intervention): This arm includes patients with intrahepatic recurrence of colorectal cancer liver metastases who underwent systemic therapy.
- systemic therapy combined with radiofrequency ablation (Experimental): This arm includes patients with intrahepatic recurrence of colorectal cancer liver metastases who underwent systemic therapy combined with radiofrequency ablation.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — This study is the first to apply radiofrequency ablation to multiple recurrent intrahepatic lesions of colorectal cancer liver metastases.
  Arms: systemic therapy combined with radiofrequency ablation

SUMMARY:
The goal of this clinical trial is to learn if radiofrequency ablation works to treat recurrent colorectal cancer liver metastases after surgery in adults. It will also learn about the safety of radiofrequency ablation. The main questions it aims to answer are:

Is radiofrequency ablation safe and effective in the treatment of recurrent colorectal cancer liver metastases? What medical problems do participants have when treating with radiofrequency ablation? Does radiofrequency ablation enable patients with recurrent colorectal cancer liver metastases to live longer? Researchers will compare systemic therapy combined with radiofrequency ablation to systemic therapy to see if radiofrequency ablation works to treat liver metastases better.

Participants will:

Receive systemic treatment for colorectal cancer liver metastases. Undergo (or not) radiofrequency ablation for colorectal cancer liver metastases.

Visit the hospital once every 3 months for checkups and tests.

DETAILED DESCRIPTION:
The percutaneous radiofrequency ablation (RFA) is guided by ultrasound imaging to target and locate the tumor, and the ablation electrode needles are inserted into the tumor foci, leading to the death of the tumor cells through direct thermal effect. In recent years, many clinical studies have confirmed that RFA is a minimally invasive, safe and effective local treatment for liver tumors, which has been widely used and studied worldwide. This study is for patients with intrahepatic multifocal recurrence after surgery for liver metastasis of colorectal cancer. Systemic therapy with/without radiofrequency ablation will be performed of intrahepatic lesions. The feasibility, efficacy and safety of the treatment strategy will be evaluated and analyzed through follow-up, which will provide a new treatment mode and a basis for clinical decision-making for patients with multiple lesions of progressive colorectal cancer.

For patients with multiple intrahepatic metastatic lesions, who are not suitable for or refuse to undergo surgical re-resection, explore the feasibility of a modality treatment of radiofrequency batch therapy combined with systemic therapy. Firstly, 2-4 cycles of systemic therapy should be performed, and the response to treatment should be evaluated by enhanced CT/MRI combined with multimodal ultrasonography, and radiofrequency ablation should be performed for patients who have effective systemic therapy. Before radiofrequency ablation treatment, relevant hematological tests, such as blood routine, biochemistry, coagulation function, etc., were performed to ensure that the enrollment criteria were met. For patients who do not meet the enrollment criteria, radiofrequency ablation treatment will be postponed and clinical treatment will be performed until the enrollment criteria are met, and those patients who cannot meet the enrollment criteria will be withdrawn from the study. Secondly, the 2-6 intrahepatic lesions for the first radiofrequency ablation were confirmed according to the ultrasound model and other clinical factors. After radiofrequency treatment, 1-2 cycles of systemic treatment were carried out, and after effective evaluation, radiofrequency ablation was performed again for 2-6 foci (the selection criteria were the same as the above), and so on, with a maximum of 3 times of ablations, to ablate all the visible foci as far as possible, and to achieve a basically no evidence of disease in the liver. Systemic therapy was separated from radiofrequency ablation therapy by 1 week to minimize the impact of treatment side effects. In the control group, patients would be treated with systemic therapy alone, without localized treatment.

Enhanced CT/MRI will be performed 1 month after radiofrequency ablation treatment to evaluate the effectiveness of the technique. Ultrasound/contrast-enhanced ultrasound imaging, enhanced CT/MRI, laboratory tests (hematology, blood biochemistry, tumor markers, etc.), electrocardiogram will be performed every 3 months within 2 years after treatment. Ultrasound/contrast-enhanced ultrasound imaging, laboratory tests, electrocardiogram will be performed every 3 months and enhanced CT/MRI every 6 months after 2 years of treatment.

Due to the large number of lesions treated with radiofrequency, the occurrence of post-radiofrequency complications is closely monitored, as well as the effect on the patient's hepatic and renal function after radiofrequency ablation. As radiofrequency ablation may reduce the times of systemic therapy, it may reduce the toxic side effects of systemic therapy. Patients in both groups were tested regularly, asked about their condition, underwent physical examination, recorded vital signs and laboratory indicators, electrocardiograms, adverse events such as drug side effects and complications of radiofrequency therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer whose primary lesions have been resected or can be controlled;
2. Multiple confined lesions in the liver, the number of which can be defined;
3. The liver contains at least 2 lesions suitable for radiofrequency ablation;
4. The maximum diameter of the intrahepatic tumor is <5 cm;
5. The location of the hepatic lesion does not show obvious invasion with neighboring organs or large blood vessels;
6. No extrahepatic metastases or stable extrahepatic metastases;
7. Re-operative hepatic surgical resection is not indicated or refused;
8. Ultrasound or ultrasonography can show intrahepatic lesions;
9. The patient and his/her family request active treatment;
10. Voluntary informed consent;
11. Male or female at least 18 years of age;
12. Platelet count >50, 000/mm3 and prothrombin activity >50%;
13. Subjects are willing to return to the study center for study follow-up;
14. Life expectancy ≥ 6 months.

Exclusion Criteria:

1. Suffering from, but not limited to, the following serious illnesses: congestive heart failure, myocardial infarction or cerebrovascular accident, or life-threatening cardiac arrhythmia within the last 6 months;
2. Pregnancy or lactation. Women of childbearing potential must have a negative serum pregnancy test prior to receiving study treatment;
3. Known hypersensitivity to any of the intravenous imaging agents that will be used in the study;
4. Have portal or hepatic vein tumor infiltration/cancer embolism;
5. Prothrombinogen international normalized ratio >1.5 times the upper limit of normal (UNL) at the study center;
6. Platelet count <50, 000/mm3, absolute neutrophil count <1500/mm3, or hemoglobin value <10.0 g/dL;
7. Serum creatinine ≥ 2.5 mg/dL or calculated creatinine clearance (CrCl) ≤ 25.0 ml/min;
8. Serum bilirubin >3.0 mg/dL;
9. Serum albumin <2.8 g/dL;
10. Body temperature >101°F (38.3°C) immediately prior to study treatment;
11. Being treated with other investigational drugs;
12. Heart failure NYHA functional class III or IV.
13. Any other circumstances that the investigator deems inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
liver progression-free survival | 2 years
  Time from initial treatment to intrahepatic disease progression or patient death

SECONDARY OUTCOMES:
overall survival | 2 years
  Time from initial treatment to patient death

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yang, PhD, Principal Investigator — Peking University Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: No